CLINICAL TRIAL: NCT05612646
Title: Taiwan Taichung Veterans General Hospital
Brief Title: The Effect of Acupressure in Improving Constipation Among Inpatients in Neurology Departments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CF20208B
Record Dates: First submitted 2022-10-25; First posted 2022-11-10 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Constipation
Keywords: acupressure, constipation,
MeSH Terms: conditions — Constipation | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: Assignment A two-group controlled, randomized study, the intervention groups: receiving acupressure on 3 acupoints (Tianshu, ST25: Stomach Meridian 25; Zhongwan CV12: Conception Vessel 12; Qihai CV6: Meridian Vessel 6), control groups: receiving routine nursing and fake acupressure.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Use the random number generator of EXCEL to generate the random number assigned by the computer, and put the serial number in the sealed envelope in sequence. After the patients completed the pre-test, the sealed envelopes were opened in sequence, and the patients were randomly assigned to the experimental group and the routine care group. The study used an assessor blinding design, that is, the data collectors were unaware of the patient group assignments until the end of the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- routine nursing and fake acupressure (Active Comparator): control groups: receiving routine nursing and fake acupressure to improve constipation for 7 days during hospitalization.
  Interventions: Procedure: routine nursing and fake acupressure
- acupressure (Experimental): The patients assigned to the experimental group received acupoint massage designed to improve constipation for 7 days during hospitalization. The selection of acupoints in this study includes "Tianshu (double)" (Tianshu, ST25: Stomach Meridian 25, the 25th point of the stomach meridian), "Zhongwan (single)" (Zhongwan CV12: Conception Vessel 12, the 12th point of the Ren meridian) ), "Qihai Point (Single)" (Qihai CV6: Meridian Vessel 6 Renmai 6th point) 3 points.
  Interventions: Procedure: Acupressure

INTERVENTIONS:
Procedure: Acupressure — The patients assigned to the experimental group received acupoint massage designed to improve constipation for 7 days during hospitalization. The selection of acupoints in this study includes "Tianshu (double)" (Tianshu, ST25: Stomach Meridian 25, the 25th point of the stomach meridian), "Zhongwan (single)" (Zhongwan CV12: Conception Vessel 12, the 12th point of the Ren meridian) ), "Qihai Point (Single)" (Qihai CV6: Meridian Vessel 6 Renmai 6th point) 3 points.
  Arms: acupressure
Procedure: routine nursing and fake acupressure — control groups: receiving routine nursing and fake acupressure to improve constipation for 7 days during hospitalization.
  Arms: routine nursing and fake acupressure

SUMMARY:
As a form of non-invasive auxiliary care, Traditional Chinese Medicine acupressure can prevent constipation, reduce medication for constipation, save medical costs, and alleviate constipation among inpatients in neurology departments, as well as improve patients' general ease and comfort of defecation, thereby improving their quality of life. It also provides clinical nursing staff with a more effective, safer, and more comfortable auxiliary method of preventing constipation, and can be used as a reference for the nursing of such patients.

DETAILED DESCRIPTION:
Background: Constipation is a common problem among geriatric patients and in neurology departments. However, using stool softeners and enemas yield only temporary effects and may even lead to alternating constipation, diarrhea, and metabolic disorders. Because of its non-invasive nature, Acupressure can be used as adjuvant therapy of integrated traditional Chinese and western medicine to prevent constipation among inpatients in neurology departments. It is necessary to verify that Acupressure can be applied to avoid and alleviate patients' constipation, improve their comfort, and improve their quality of life.

Objective: To explore the effect of Acupressure in alleviating constipation among inpatients in neurology departments.Method: A randomized controlled two-group pre-test and post-test experiment design were adopted in this study; neurology department inpatients were randomly assigned to either the experimental group, which comprised 64 subjects receiving Acupressure on three acupoints (Tianshu, ST25: Stomach Meridian 25; Zhongwan CV12: Conception Vessel 12; Qihai CV6: Meridian Vessel 6) or the control group which comprised 64 subjects receiving routine nursing and fake Acupressure. The research tools included the Bristol Stool Form and Constipation Assessment Scale.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 20 years old
2. Established diagnosis of stroke (ischemic, hemorrhagic acute phase)
3. NIHSS 1-20 points
4. Undiagnosed within three months before admission With intestinal disease and no rectal resection
5. meeting the diagnostic criteria for functional constipation (Rome IV).

Exclusion Criteria:

1. Abdominal surgery or abdominal radiotherapy within three months
2. Abdominal cancer including liver, large intestine, lymph, and pelvic cavity, etc.,
3. Massive ascites
4. There are implants in the abdominal cavity, such as V-P Shunt, L-P Shunt, CAPD, etc.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 128 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
The constipation assessment scale scores | Assessment from the first day to the seventh day after treatment
  Constipation Assessment Scale (CAS), a total of 8 questions, 0 points: no, 1 point: yes, but not severe, 2 points. Very serious, the higher the score (0-16 points), the more severe the constipation symptoms.
The Bristol Stool Form Scale | Assessment from the first day to the seventh day after treatment
  bach's alpha of The Bristol Stool Form Scale. Classification: Type 1: hard balls (difficult to pass through), Type 2: sausage-like, but with uneven surface Type 3: sausage-like, but with cracks on the surface, Type 4: like sausage or snake Surface is smooth, type 5: soft lumps with smooth broken edges (easy to pass), type 6: fluffy lumps with rough edges, mushy stool, type 7: watery, no solid lumps (completely liquid), type 1 Types 3 and 2 indicate constipation; Types 3 and 4 are ideal stool shapes, especially Type 4 is the easiest to defecate; Types 5 to 7 are likely to have diarrhea

CONTACTS AND LOCATIONS:
Overall Officials: Hsiao-Chi Nieh, MSC, Study Chair — Head Nurse
Locations (1):
- 1650 Taiwan Boulevard Sect. 4, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abbasi P, Mojalli M, Kianmehr M, Zamani S. Effect of acupressure on constipation in patients undergoing hemodialysis: A randomized double-blind controlled clinical trial. Avicenna J Phytomed. 2019 Jan-Feb;9(1):84-91. PMID 30788281
- [Result] Bharucha AE, Lacy BE. Mechanisms, Evaluation, and Management of Chronic Constipation. Gastroenterology. 2020 Apr;158(5):1232-1249.e3. doi: 10.1053/j.gastro.2019.12.034. Epub 2020 Jan 13. PMID 31945360
- [Result] Birimoglu Okuyan C, Bilgili N. Effect of abdominal massage on constipation and quality of life in older adults: A randomized controlled trial. Complement Ther Med. 2019 Dec;47:102219. doi: 10.1016/j.ctim.2019.102219. Epub 2019 Oct 16. PMID 31780015
- [Result] Chen MC, Yang LY, Chen KM, Hsu HF. Systematic Review and Meta-Analysis on Using Acupressure to Promote the Health of Older Adults. J Appl Gerontol. 2020 Oct;39(10):1144-1152. doi: 10.1177/0733464819870027. Epub 2019 Aug 19. PMID 31426687
- [Result] Chumpitazi BP, Self MM, Czyzewski DI, Cejka S, Swank PR, Shulman RJ. Bristol Stool Form Scale reliability and agreement decreases when determining Rome III stool form designations. Neurogastroenterol Motil. 2016 Mar;28(3):443-8. doi: 10.1111/nmo.12738. Epub 2015 Dec 21. PMID 26690980
- [Derived] Nieh HC, Wu PO, Ou SF, Li HP, Chen JP. Effect of acupressure on alleviating constipation among inpatients with stroke during the acute phase: A randomized controlled trial. Complement Ther Clin Pract. 2023 Nov;53:101801. doi: 10.1016/j.ctcp.2023.101801. Epub 2023 Sep 22. PMID 37793306